CLINICAL TRIAL: NCT00564122
Title: A Comparison of the Accuracy of an Artificially-Intelligent Stethoscope Versus Pediatric Cardiologists in the Assessment of Pediatric Patients Referred to a Cardiologist for the Assessment of a Heart Murmur
Brief Title: The Accuracy of an Artificially-intelligent Stethoscope
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Collaborators: Thomas C. Dispenza, M.D. (Unknown); John R. Bockoven, M.D. M.B.A. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 070904
Record Dates: First submitted 2007-11-23; First posted 2007-11-27 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Heart Murmurs; Congenital Heart Disease; Structural Heart Disease
Keywords: Murmur; Artificial-Intelligence; Stethoscope; Congenital Heart Disease; Structural Heart Disease
MeSH Terms: conditions — Heart Murmurs; Heart Defects, Congenital | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All subjects
  Interventions: Device: Artificially-Intelligent Stethoscope; Other: Physical Examination

INTERVENTIONS:
Device: Artificially-Intelligent Stethoscope — After subjects' medical visits are complete, the heart sounds of all subjects will be recorded and assessed by an artificially-intelligent stethoscope. Attempts will be made to make satisfactory 20-second recordings from a total of eight positions on the chest with the patient in supine and upright positions.
  Other Names: Cardioscan, Zargis Medical Corporation, Serial Number 000127
Other: Physical Examination — A Pediatric Cardiologist will examine each subject to the extent needed to make clinical assessments. This represents the ordinary standard-of-care.

SUMMARY:
This study will characterize the accuracy of a commercially available artificially-intelligent stethoscope in determining which childhood murmurs suggest underlying congenital structural heart disease and therefore warrant diagnostic echocardiograms.

DETAILED DESCRIPTION:
Heart murmurs can be ausculted in most pediatric patients, but underlying Congenital Structural Heart (CSH) Disease is rare. Nevertheless, CSH Disease is often first suggested by the presence of a murmur. Primary care providers refer pediatric patients to Cardiologists for murmur evaluations with low accuracy, and this pattern results in:

1. needless emotional strain on many patients with functionally normal hearts and their families,
2. increased morbidity and mortality rates for rare patients with delayed cardiac diagnoses, and
3. exorbitant costs to society.

Referral accuracy for murmur evaluations probably is low because the differences between innocent and pathological murmurs can be subtle. Computer-assisted analysis of heart sounds may increase the accuracy of primary care referrals to pediatric cardiologists, but the accuracy of the only FDA-approved artificially-intelligent cardiac auscultation system, Zargis Medical Corporation's Cardioscan®, has never been determined prospectively in an unselected population of live pediatric patients. As a primary endpoint, the study herein proposed would prospectively compare the sensitivity and specificity of the Cardioscan® with that of CHMCA's Pediatric Cardiologists in the identification of cardiac pathology among 300 new and unselected pediatric patients referred to CHMCA's cardiologists for murmur evaluations, using two-dimensional transthoracic echocardiography as the common gold-standard. Double-blinding will be in place. The study also will attempt secondarily to gauge the clinical significance of pathology missed by the Cardioscan®, to define sub-populations of patients among which the Cardioscan's® judgment should be considered less accurate, and to gather data concerning the value and acceptability to families of the Cardioscan®. If (as expected) the Cardioscan's® accuracy merely approaches that of Pediatric Cardiologists, then the study herein proposed would still establish the Cardioscan® as a formidable tool for primary care providers-a helpful, billable, and potentially cost-saving alternative to consulting Cardiology on patients with probably- or possibly-innocent murmurs. Data collection for this project will occur predominantly within CHMCA's Heart Center in Akron, although some data collection may occur within CHMCA and/or at CHMCA's Heart Centers in Beachwood and/or Boardman. Minimal disruption to existing clinical patient flow through those settings would be expected and the entire protocol is expected to be completely painless and noninvasive, with no foreseeable health risks.

ELIGIBILITY:
Inclusion Criteria:

* The patient must present to a consulted cardiologist for a 1st non-primary care murmur evaluation.

Exclusion Criteria:

* Non English-speakers
* At least moderately agitated or disruptive patients
* An echocardiogram or a Cardiology evaluation was done previously
* The patient no longer has an ausculable murmur at presentation.
* The patient didn't have a transthoracic echocardiogram with Color Doppler done.
* Patients admitted to the NICU before protocol completes.
* Protocol can't be completed on the day of presentation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient must present to a consulted Cardiologist for a 1st non-primary care murmur evaluation. This will usually occur in an outpatient Pediatric Cardiology clinic site.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-12; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the Artificially-Intelligent Stethoscope as compared with that of Pediatric Cardiologists in determining which patients needed echocardiograms because they have congenital structural heart disease | Not applicable; all data collection for any given patient will be completed within less than 12 hours--usually MUCH less than 12 hours.

SECONDARY OUTCOMES:
Specificity of the Artificially-Intelligent Stethoscope as compared with that of Pediatric Cardiologists in determining which patients needed echocardiograms because they have congenital structural heart disease. | Not applicable; all data collection for any given patient will be completed within less than 12 hours--usually MUCH less than 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Dispenza, M.D., Principal Investigator — Akron Children's Hospital; John R. Bockoven, M.D. M.B.A., Principal Investigator — Akron Children's Hospital
Locations (3):
- United States (3):
  - Akron Children's Hospital's Heart Center, Akron, Ohio
  - Akron Children's Hospital's Heart Center, Beachwood, Ohio
  - Akron Children's Hospital's Heart Center, Boardman, Ohio